CLINICAL TRIAL: NCT03328156
Title: Erectile Dysfunction After Percutaneous Coronary Intervention Versus the Thrombolytic Therapy in Acute ST Elevation Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Mahmmoud Syed, Cardiology Resident, Assiut University
Other Study IDs: 17100377
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with STEMI will treated by PPCI: Primary angioplasty procedure The procedure will be performed using a standard angioplasty technique. A bolus of100 IU kg of heparin will be administered intra-arterially after insertion of the vascular catheter. The target lesions will initially treated with appropriate balloon predilatation as necessary, followed by intracoronary stenting. After stent implantation, heparin will be routinely administered. The sheaths will be removed the same day.
- patient with STEMI will treated by Thrombolytic therapy: oral clopidogrel (300 mg), Low-flow nasal oxygen, oral acetylsalicylic acid (325 mg), Will be given to each patient. Streptokinase will be given intravenously at 1.5 million units over approximately 60 min. Reperfusion afterTT will be assessed according to clinical criteria .

SUMMARY:
Erectile dysfunction is a common sexual problem affecting up to one-third of men throughout their life. It is now well recognized that risk factors for erectile dysfunction (ED) include the same risk factors as coronary artery disease, including smoking, dyslipidemia, diabetes, hypertension, lack of physical activity and obesity. We will investigate the effect of reperfusion strategies (primary angioplasty & therapeutic therapy) on the prevalence of erectile dysfunction after acute myocardial infarction. Erectile function will be evaluated using the international index of erectile function after 3 months of successful reperfusion treatment of acute myocardial infarction.

DETAILED DESCRIPTION:
Myocardial infarction the term acute myocardial infarction(AMI) should be used when there is evidence of myocardial injury (defined as an elevation of cardiac troponin values with at least one value above the 99th percentile upper reference limit) with necrosis in a clinical setting consistent with myocardial ischemia . Myocardial infarction is classified as either : ST elevation acute myocardial infarction.* non-ST segment elevation acute myocardial infarction. according to the electrocardiogram at the time of admission.

There are Two main treatment modalities for STEMI which are primary percutaneous coronary intervention (PPCI) & thrombolytic treatment (TT).

* Erectile dysfunction (ED) is defined as the recurrent or persistent inability to achieve and/or maintain an erection for satisfactory intercourse.Erectile function will be evaluated using the international index of erectile function in the hospital to characterize each patients sexual function before the acute myocardial infarction & 3 months after the event.

International Index of Erectile Function (IIEF-5) Questionnaire

1. How do you rate your confidence that could you get and keep an erection? 1)very low 2)low 3)moderate 4)high 5)very high
2. . When you had erections with sexual stimulation, how often were your erections hard enough for penetration?

1) Almost never/never 2) A few times (much less than half the time) 3) Sometimes (about half the time) 4) Most times (much more than half the time) 5) Almost always/always 3-During sexual intercourse, how often were you able to maintain your erection after you had penetrated (entered) your partner?

1. Almost never/never
2. A few times (much less than half the time)
3. Sometimes (about half the time)
4. Most times (much more than half the time)
5. Almost always/always 4- During sexual intercourse, how difficult was it to maintain your erection to completion of intercourse?

1) Extremely difficult 2) Very difficult 3) Difficult 4) Slightly difficult 5) Not difficult 5- When you attempted sexual intercourse, how often was it satisfactory for you?

1. ) Almost never/never
2. A few times (much less than half the time)
3. Sometimes (about half the time)
4. Most times (much more than half the time)
5. Almost always/always the cases will be classified as:

   * without ED (score greater than 25 points)
   * mild ED (score 17 to 25),
   * moderate ED (score 11 to 16)
   * severe ED (score 10 points or less). No treatment for ED would applied within the 3-month period prior to the second IIEF evaluation for each patient

ELIGIBILITY:
Inclusion Criteria:

* patients with ST elevation myocardial infarction undergo to of successful reperfusion treatment

Exclusion Criteria:

* - patients with an atrial fibrillation or flutter.
* -patients who cannot be reperfused with thrombolytic therapy and require emergency percutaneous coronary intervention (causing crossover between the groups).
* congenital disease
* pericardial disease
* patients with renal failure
* severe valvular heart disease
* liver cirrhosis
* thyroid disease
* previous pelvic, penile, urethral or prostate surgery

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In this study; we aim to investigate the effects of two different reperfusion strategies (primary angioplasty & therapeutic therapy) on the prevalence of erectile dysfunction after acute myocardial infarction.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
The International Index of Erectile Function (IIEF-5) Questionnaire | 3 months
  the cases will be classified as:
  * without ED (score greater than 25 points)
  * mild ED (score 17 to 25),
  * moderate ED (score 11 to 16)
  * severe ED (score 10 points or less). No treatment for ED would applied within the 3-month period prior to the second IIEF evaluation for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Taha Keshk, MD, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Lewis RW. A critical look at descriptive epidemiology of sexual dysfunction in Asia compared to the rest of the world - a call for evidence-based data. Transl Androl Urol. 2013 Mar;2(1):54-60. doi: 10.3978/j.issn.2223-4683.2013.01.03. PMID 26816724
- [Background] Hellstrom WJ. Does erectile dysfunction drug use contribute to risky sexual behavior? Asian J Androl. 2010 Sep;12(5):626-7. doi: 10.1038/aja.2010.98. No abstract available. PMID 20818401
- [Background] Montorsi P, Montorsi F, Schulman CC. Is erectile dysfunction the "tip of the iceberg" of a systemic vascular disorder? Eur Urol. 2003 Sep;44(3):352-4. doi: 10.1016/s0302-2838(03)00307-5. No abstract available. PMID 12932935
- [Background] O'Kane PD, Jackson G. Erectile dysfunction: is there silent obstructive coronary artery disease? Int J Clin Pract. 2001 Apr;55(3):219-20. PMID 11351777
- [Background] Borgquist R, Gudmundsson P, Winter R, Nilsson P, Willenheimer R. Erectile dysfunction in healthy subjects predicts reduced coronary flow velocity reserve. Int J Cardiol. 2006 Sep 20;112(2):166-70. doi: 10.1016/j.ijcard.2005.08.035. Epub 2005 Nov 4. PMID 16271777
- [Background] Ho CC, Singam P, Hong GE, Zainuddin ZM. Male sexual dysfunction in Asia. Asian J Androl. 2011 Jul;13(4):537-42. doi: 10.1038/aja.2010.135. Epub 2011 Jun 6. PMID 21643001
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction; Jaffe AS, Apple FS, Galvani M, Katus HA, Newby LK, Ravkilde J, Chaitman B, Clemmensen PM, Dellborg M, Hod H, Porela P, Underwood R, Bax JJ, Beller GA, Bonow R, Van der Wall EE, Bassand JP, Wijns W, Ferguson TB, Steg PG, Uretsky BF, Williams DO, Armstrong PW, Antman EM, Fox KA, Hamm CW, Ohman EM, Simoons ML, Poole-Wilson PA, Gurfinkel EP, Lopez-Sendon JL, Pais P, Mendis S, Zhu JR, Wallentin LC, Fernandez-Aviles F, Fox KM, Parkhomenko AN, Priori SG, Tendera M, Voipio-Pulkki LM, Vahanian A, Camm AJ, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Morais J, Brener S, Harrington R, Morrow D, Lim M, Martinez-Rios MA, Steinhubl S, Levine GN, Gibler WB, Goff D, Tubaro M, Dudek D, Al-Attar N. Universal definition of myocardial infarction. Circulation. 2007 Nov 27;116(22):2634-53. doi: 10.1161/CIRCULATIONAHA.107.187397. Epub 2007 Oct 19. No abstract available. PMID 17951284
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Greenstein A, Chen J, Miller H, Matzkin H, Villa Y, Braf Z. Does severity of ischemic coronary disease correlate with erectile function? Int J Impot Res. 1997 Sep;9(3):123-6. doi: 10.1038/sj.ijir.3900282. PMID 9315488
- [Background] Chughtai B, Lee RK, Te AE, Kaplan SA. Metabolic syndrome and sexual dysfunction. Curr Opin Urol. 2011 Nov;21(6):514-8. doi: 10.1097/MOU.0b013e32834b8681. PMID 21897258
- [Background] Jackson G, Solomon H, Wierzbicki AS. Letter regarding article by Gazzaruso et al, "Relationship between erectile dysfunction and silent myocardial ischemia in apparently uncomplicated, type 2 diabetic patients". Circulation. 2005 Jan 18;111(2):e18-9; author reply e18-9. doi: 10.1161/01.CIR.0000152482.71628.51. No abstract available. PMID 15657383